CLINICAL TRIAL: NCT00156052
Title: A Randomized Trial of Hypofractionated Radiotherapy Post-Lumpectomy in Women With Node Negative Breast Cancer
Brief Title: Hypofractionated Radiotherapy Post-Lumpectomy in Women With Node Negative Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCOG-1993-hypo
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Hypofractionated Radiotherapy; Lumpectomy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypofractionated whole breast radiation (Experimental): Subjects treated with 4250 cGY in 16 fractions
  Interventions: Radiation: Hypofractionated whole breast radiation schedule
- Conventional whole breast radiation (Active Comparator): Subjects treated with 5000 cGY in 25 fractions
  Interventions: Radiation: Conventional whole breast radiation schedule

INTERVENTIONS:
Radiation: Conventional whole breast radiation schedule
  Arms: Conventional whole breast radiation
Radiation: Hypofractionated whole breast radiation schedule
  Arms: Hypofractionated whole breast radiation

SUMMARY:
To determine if hypofractionated radiotherapy to the whole breast (4,250 cGy/16 fractions over 22 days) is equally effective to standard fractionated radiotherapy (5,000 cGy/25 fractions over 35 days) in women with node negative breast cancer who have undergone lumpectomy.

The primary outcome is local breast recurrence and secondary outcomes include morbidity and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. The female patient has a histological diagnosis of invasive carcinoma of the breast, and no evidence of metastatic disease.
2. Has had a lumpectomy (including segmental resection and partial mastectomy), that is, surgical excision of the tumour with a rim of normal tissue.
3. Patient has not had an axillary dissection, OR for patients who have had an axillary dissection, all nodes are negative for metastatic disease.

Exclusion Criteria:

1. Tumour greater than 5 cm in greatest diameter on pathological examination.
2. The presence of invasive or intraductal (noninvasive) breast cancer involving the surgical margins.
3. Clinical evidence prior to surgery of infiltration of the skin of the involved breast such as edema, ulceration, or fixation of the tumour to underlying muscle, or inflammatory breast cancer.
4. Bilateral malignancy of the breast (synchronous or metachronous).
5. More than one primary invasive tumour in the same breast.
6. Previous surgery for breast cancer.
7. Pathological status of axilla is unknown.
8. Status for adjuvant systemic therapy not determined.
9. For patients not treated with adjuvant chemotherapy: unable to commence radiation therapy within 16 weeks of last surgical procedure on the breast.
10. For patients treated with adjuvant chemotherapy: unable to commence radiation therapy within 8 weeks of the last dose of chemotherapy.
11. Serious nonmalignant disease (eg. cardiovascular, renal, etc.) which would preclude surgical or radiation treatment.
12. Currently pregnant or lactating.
13. Breast deemed too large to permit satisfactory radiation (ie. separation > 25 cm).
14. Previous concomitant malignancies of any type except squamous, or basal cell carcinomas of the skin, or carcinoma \fIin situ\fR of the cervix which have been effectively treated.
15. Geographic inaccessibility for follow-up.
16. Psychiatric or addictive disorders which preclude obtaining informed consent or adherence to the protocol.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1234 (Actual)
Dates: Start 1993-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Local breast recurrence | Indefinitely

SECONDARY OUTCOMES:
Morbidity | Indefinitely
Cost effectiveness | Indefinitely

CONTACTS AND LOCATIONS:
Overall Officials: Tim Whelan, MD, Study Chair — Juravinski Cancer Centre
Locations (11):
- Canada (11):
  - Regional Cancer Program of the Sudbury Regional Hospital, Greater Sudbury, Ontario
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Centre, London, Ontario
  - Ottawa Hospital-Integrated Cancer Program, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Regional Cancer Care - Thunder Bay HSC, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - The Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - Montreal General Hospital, Montreal, Quebec

REFERENCES:
- [Result] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639
- [Result] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717